CLINICAL TRIAL: NCT03676751
Title: Gut and Azithromycin Mechanisms in Infants and Neonates
Brief Title: MORDOR II Burkina Faso: Longitudinal Trial
Acronym: GAMIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OPP1187628-C
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Child Growth; Diversity of Microbiome; Child Mortality; Resistance Bacterial
Keywords: azithromycin; mass drug administration; childhood mortality
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Individually randomized placebo-controlled trail of azithromycin vs. placebo to establish the efficacy and safety of azithromycin.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Active Comparator): A single dose of azithromycin will be administered to children between the ages of 8 days and 59 months old.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): A single dose of placebo will be administered to children between the ages of 8 days and 59 months old.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Zithromax® for oral suspension is supplied in bottles containing azithromycin dehydrate powder equivalent to 1200mg per bottle and the following inactive ingredients: sucrose; tribasic anhydrous sodium phosphate; hydroxypropyl cellulose; xanthan gum; FD&C Red #40; and flavoring including spray dried artificial cherry, crème de vanilla, and banana. After constitution, a 5mL suspension contains 200mg of azithromycin.
  Arms: Azithromycin
Drug: Placebo — Oral suspension of placebo for azithromycin
  Arms: Placebo

SUMMARY:
Globally, childhood mortality has shown a promising downward trend in recent years, however, many sub-Saharan countries still have relatively high child mortality rates. In previous studies within Niger, Tanzania, and Malawi, mass azithromycin treatment to children aged 1-59 months old effectively reduced all-cause childhood mortality. A similar study will be conducted in Burkina Faso to replicate the results of mass azithromycin treatment.

The investigators propose an individually randomized placebo-controlled trial alongside the MORDOR II Burkina Faso trial to evaluate the effect of a single dose of azithromycin (20 mg/kg) on potential mediators of the effect of azithromycin on all-cause mortality. Many questions surround the mechanism behind azithromycin's effect on reducing childhood mortality. Further questions exist regarding antibiotic resistance and how mass antibiotic administration can impact intestinal microflora. The goal of this study is to demonstrate the changes in the gut microbiome after antibiotic administration and to measure the growth of children after receiving a single dose of azithromycin. Additionally we will measure resistance markers, inflammatory markers, and IgA-bound bacteria. We hypothesize that a single dose of azithromycin will lead to a significant increase in child growth and that the gut microbiome will be significantly different in children who received azithromycin compared to those who received placebo.

Objectives:

1. . To determine the effect of a single dose of azithromycin for children aged 8 days-59 months on longitudinal changes in the intestinal microbiome over a 6-month period. We hypothesize that a single dose of azithromycin will result in a significant difference in the intestinal microbiome within the treatment group compared to the placebo group after a 6-month period within children ages 8 days-59 months.
2. . To determine the effect of a single dose of azithromycin for children aged 8 days-59 months on child growth over a 6-month period. We hypothesize that a single dose of azithromycin will increase child growth over a 6-month period in children aged 8 days-59 months.
3. . To determine the effect of a single dose of azithromycin for children aged 8 days to 59 months on the presence of macrolide genetic resistance determinants within the first two weeks post-treatment. The investigators hypothesize that a single dose of azithromycin will increase the presence of macrolide resistance determinants over a 2 week period in children aged 8 days to 59 months.

The study will be conducted in Nouna Town in northwestern Burkina Faso.

DETAILED DESCRIPTION:
The investigators' previous MORDOR I research demonstrated a significant reduction in all-cause child mortality after biannual mass azithromycin distribution. In three sub-Saharan Africa countries, (including Niger, Tanzania, and Malawi) mass azithromycin treatment over 2 years resulted in a 14% reduction in child mortality. Moreover, 1 in 5-6 deaths were shown to be averted within Niger alone1. Similar findings were demonstrated in a previous study for trachoma control in Ethiopia with mass azithromycin distribution. This study in rural Ethiopia noted a nearly 50% decrease in all-cause childhood mortality5. However, neither of these studies evaluated the longitudinal impact azithromycin has on the gut microbiome. The MORDOR II trial in Burkina Faso will further evaluate the efficacy of biannual azithromycin treatment. The under-5 child mortality rate in Burkina Faso is approximately 110 per 1,000 live births. Major causes of child mortality in this area are infectious mostly due to malaria, diarrhea, and upper respiratory tract infections. In addition, malnutrition contributes to a high burden of child mortality and morbidity within this region as well. By treating underlying conditions, the use of routine antibiotic treatment could reduce diverse health outcomes leading to morbidity and mortality. The investigative team proposes to conduct this study alongside the MORDOR II trial in the town of Nouna where a majority of childhood deaths are attributable to infectious causes and malnutrition.

The World Health Organization is considering adopting the presumptive use of azithromycin and other antibiotics as a recommendation to reduce childhood mortality in areas with a high infectious disease burden2. Many questions remain unanswered surrounding the use of mass antibiotic treatment in areas with high child morbidity and mortality. This study will add to the current knowledge of mass azithromycin distribution from our previous MORDOR I research. The investigators propose to evaluate how azithromycin will impact childhood growth and to assess the changes that occur in the intestinal microbiome following a single dose of azithromycin treatment. The goal is to contribute more scientific literature that could assist future guidelines regarding antibiotic use.

The role of antibiotics on child growth is unclear. Recent studies indicate that antibiotic use could impact child growth, but a previous study in Niger failed to find a statistically significant correlation between antibiotic treatment with azithromycin and stunting, underweight, or MUAC of pre-school aged children. Longitudinal studies have been recommended to further investigate the role of antibiotics on child growth6. Meanwhile some studies suggest antibiotics may create modifications in the gut microbiota impacting nutrient absorption and weight gain7.The investigative team proposes to measure child growth through anthropometric measurements longitudinally over a 6-month period to see if azithromycin treatment impacts child development. We hypothesize that children receiving a dose of azithromycin will have more growth and development in terms of height, weight, and mid-upper arm circumference compared to children who receive placebo.

The investigators propose a longitudinal study designed to improve our knowledge about the changes in the intestinal microbiome following the course of a single dose of antibiotic in a setting with high childhood mortality and morbidity. More specifically, we propose to follow 500 children for a 6-month time period that are between the ages of 8 days old and 59 months old. Children in this age bracket are at the highest risk for mortality from infectious causes, and furthermore, they are at the highest risk for malnutrition. This group of children would receive the greatest benefit from this intervention. The causal changes in the microbiome are vastly understudied in regards to changes in the gut microbiome following a course of antibiotics. The investigators hypothesize that children receiving a dose of azithromycin will have a higher prevalence of pneumococcal resistance in nasopharyngeal samples, decreased bacterial diversity, and a higher likelihood of identification of bacterial resistance genes in stool and nasopharyngeal samples.

A small group of 50 children (25 per arm) will be followed more intensely within the first 2 weeks of treatment to evaluate macrolide resistance. The investigators hypothesize that children receiving azithromycin will have a greater presence of macrolide genetic resistant determinants.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 days and 59 months old
* Primary residence within catchment area of study site
* Available for full 6 month study
* No known allergy to macrolides/azalides
* Appropriate written informed consent from at least one parent or guardian
* Able to feed orally

Exclusion Criteria:

* <8 days old or >59 months
* Primary residence outside catchment area of study site
* Not available for full 6 month study
* Known allergy to macrolides/azalides
* No written informed consent from at least one parent or guardian
* Unable to feed orally

Ages: 8 Days to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, PhD, Principal Investigator — University of California, San Francisco; Ali Sie, MD, PhD, Principal Investigator — Centre de Recherce en Sante de Nouna; Tom Lietman, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Centre de Recherche en Sante de Nouna, Nouna, Burkina Faso

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doan T, Liu Z, Sie A, Dah C, Bountogo M, Ouattara M, Coulibaly B, Kiemde D, Zonou G, Nebie E, Brogdon J, Lebas E, Hinterwirth A, Zhong L, Chen C, Zhou Z, Porco T, Arnold BF, Oldenburg CE, Lietman TM. Gut Microbiome Diversity and Antimicrobial Resistance After a Single Dose of Oral Azithromycin in Children: A Randomized Placebo-Controlled Trial. Am J Trop Med Hyg. 2024 Jan 16;110(2):291-294. doi: 10.4269/ajtmh.23-0651. Print 2024 Feb 7. PMID 38227963
- [Derived] Coulibaly B, Kiemde D, Zonou G, Sie A, Dah C, Bountogo M, Brogdon J, Hu H, Lebas E, Porco TC, Doan T, Lietman TM, Oldenburg CE. Effect of Single-dose Azithromycin on Pneumococcal Carriage and Resistance: A Randomized Controlled Trial. Pediatr Infect Dis J. 2022 Sep 1;41(9):728-730. doi: 10.1097/INF.0000000000003585. Epub 2022 May 23. PMID 35944061
- [Derived] Coulibaly B, Sie A, Dah C, Bountogo M, Ouattara M, Compaore A, Nikiema M, Tiansi JN, Sibiri ND, Brogdon JM, Lebas E, Doan T, Porco TC, Lietman TM, Oldenburg CE. Effect of a single dose of oral azithromycin on malaria parasitaemia in children: a randomized controlled trial. Malar J. 2021 Aug 31;20(1):360. doi: 10.1186/s12936-021-03895-9. PMID 34465327
- [Derived] Sie A, Coulibaly B, Dah C, Bountogo M, Ouattara M, Compaore G, Brogdon JM, Godwin WW, Lebas E, Doan T, Arnold BF, Porco TC, Lietman TM, Oldenburg CE. Single-dose azithromycin for child growth in Burkina Faso: a randomized controlled trial. BMC Pediatr. 2021 Mar 17;21(1):130. doi: 10.1186/s12887-021-02601-7. PMID 33731058

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 230 | 220
Received Allocated Treatment | 227 | 214
Week 14 Follow up | 218 | 203
Completed (Month 6) | 200 | 189
Not Completed | 30 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 230 | 220 | 450
Age, Continuous [Mean (Inter-Quartile Range); unit: months] | 28 [15 to 39] | 28 [17 to 38] | 28 [16 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 106 | 228
  Male | 108 | 114 | 222
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 230 | 220 | 450
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Burkina Faso | 230 | 220 | 450
Mother's age [Mean (Inter-Quartile Range); unit: years] | 28 [23 to 32] | 28 [23 to 33] | 28 [23 to 33]
Mother's education [Count of Participants; unit: Participants]
  None | 120 | 122 | 242
  Primary | 61 | 56 | 117
  Secondary or higher | 49 | 42 | 91
Mid-upper arm circumference, cm [Mean (Inter-Quartile Range); unit: cm] | 14.1 [13 to 15] | 14.4 [13.5 to 15] | 14.3 [13.5 to 15]
Weight, kg [Mean (Inter-Quartile Range); unit: kg] | 11.2 [8.8 to 13.5] | 11.5 [9.4 to 13.4] | 11.4 [9.0 to 13.4]
Height, cm [Mean (Standard Deviation); unit: cm] | 85.3 (12.2) | 85.4 (11.8) | 85.4 (12.0)
Weight-for-height Z-score [Mean (Standard Deviation); unit: score] — Nutritional status as determined by weight-for-height Z-score vs. Placebo household Weight-for-height Z-score in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Weight-for-height Z (WHZ) scores were calculated based on the 2006 World Health Organization (WHO) standards. The mean of the 2006 population standards is 0. Lower standard deviations = worse outcomes. A cutoff of < -2 means moderately wasted (WHZ). A cutoff of < -3 means wasted (WHZ).
  score | -0.6 (1.2) | -0.4 (1.1) | -0.5 (1.2)
Height-for-age Z-score [Mean (Standard Deviation); unit: score] — Nutritional status as determined by height-for-age Z-score Height-for-age Z-score in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Height-for-age Z (HAZ) score were calculated based on the 2006 World Health Organization (WHO) standards. The mean of the 2006 population standards is 0. Lower standard deviations = worse outcomes. A cutoff of < -2 means moderately stunted (HAZ). A cutoff of < -3 means severely stunted (HAZ).
  score | -0.9 (1.3) | -0.8 (1.3) | -0.9 (1.3)
Weight-for-age Z-score [Mean (Standard Deviation); unit: score] — Nutritional status as determined by weight-for-age Z-score vs. Placebo household Weight-for-age Z-score in each antibiotic group compared with placebo 4 weeks after last antibiotic dose Weight-for-age Z-score (WAZ) scores were calculated based on the 2006 World Health Organization (WHO) standards. The mean of the 2006 population standards is 0. Lower standard deviations = worse outcomes. A cutoff of < -2 means moderately underweight (WAZ). A cutoff of < -3 means severely underweight (WAZ).
  score | -1.0 (1.1) | -0.7 (1.1) | -0.9 (1.1)
Wasted (WHZ < -2) [Count of Participants; unit: Participants] | 25 | 13 | 38
Stunted (HAZ < -2) [Count of Participants; unit: Participants] | 35 | 25 | 60
Underweight (WAZ < -2) [Count of Participants; unit: Participants] | 42 | 20 | 62
Mid-upper arm circumference < 12.5 cm [Count of Participants; unit: Participants] | 11 | 7 | 18
Malaria RDT Positive [Count of Participants; unit: Participants] | 14 | 8 | 22

OUTCOME MEASURES:

1. Primary Outcome: Intestinal Microbial Diversity
Description: The primary outcome of the study was pre-specified as α-diversity (inverse Simpson's) at the genus level, expressed in effective number. The minimum of Simpson's index of diversity is 0, there is no maximum. Higher Simpson's index of diversity means more diverse. There are no subscales.
Time Frame: 6 months
Population: Analysis was done 5-pooled.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 200 | 191
index score | 46.3 (9.4) | 49.5 (11.8)

2. Primary Outcome: Macrolide Resistance
Description: Presence of macrolide genetic resistance determinants measured using DNA-seq from rectal swabs from 450 children.
  Macrolide resistance is defined by resistance to erythromycin or clarithromycin.
  We compare the read numbers of macrolide resistance in each treatment group. A higher read number indicates more resistance.
Time Frame: 2 weeks
Population: We were able to follow up with 221 patients in the azithromycin arm and 208 children in the placebo arm.
Measure: Mean (Standard Deviation); unit: number of reads
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 208
number of reads | 98.89 (184.62) | 0.5 (3.24)

3. Secondary Outcome: Change in Weight Over Time
Description: WAZ. Weight will be measured at all follow-ups and weight-for-age z-scores will be calculated. Weight measured in kg.
Time Frame: 180 days post-treatment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 218 | 203
kg | 12.5 (3.0) | 12.6 (2.8)

4. Secondary Outcome: Change in Height Over Time
Description: Height or length will be measured at all follow-ups and height-for-age z-scores will be calculated.
Time Frame: 180 days post-treatment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 200 | 189
cm | 91.6 (11.5) | 91.3 (10.6)

5. Secondary Outcome: Number of Participants With Infantile Hypertrophic Pyloric Stenosis
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 185 | 177
Participants | 0 | 0

6. Secondary Outcome: Mortality
Description: Vital status will be assessed at all follow-up time points. Mortality will be defined as death within the study period. Date of death will be collected.
Time Frame: 180 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 185 | 177
Participants | 0 | 0

7. Secondary Outcome: Malaria Status
Description: Number of Participants Positive for Malaria. Blood smears (thin and thick) for malaria will be collected at all follow-ups to determine malaria infection status.
Time Frame: 180 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 185 | 177
Participants | 14 | 10

8. Secondary Outcome: Adverse Events
Description: Caregivers will be asked if the child has been taken to the health post since the last visit and why
Time Frame: 14 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 209
Participants | 44 | 42

9. Secondary Outcome: Genotypic Resistance
Description: Total resistance read numbers in 12 classes: Aminoglycosides, Cationic antimicrobial peptides, Elfamycins, MLS, Metronidazole, Multi-drug resistance, Phenicol, Rifampin, Sulfonamides, Tetracyclines, Trimethoprim, and Beta-lactams.
  We compare the read numbers of macrolide resistance in each treatment group. A higher read number indicates more resistance.
Time Frame: 180 days post-treatment
Population: We were able to follow up with 200 children in the azithromycin group and 191 children in the placebo group.
Measure: Number; unit: number of reads
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 200 | 191
number of reads | 7547 | 13077

10. Secondary Outcome: Inflammatory Marker Changes
Description: Measured by C-reactive protein
Time Frame: 6 months
Population: The Inflammatory marker changes data is not collected in this study
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: IgA-bound Bacteria From Small Intestine Changes
Description: Measured using BugFACS from whole blood and stool
Time Frame: 180 days post-treatment
Population: Data is not collected
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Nutritional Status
Description: To be measured using mid-upper arm circumference
Time Frame: 180 days post-treatment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 200 | 189
cm | 14.3 (1.2) | 14.5 (1.0)

13. Secondary Outcome: Acute Modulation of the Gut Microbiome
Description: Next generation sequencing
Time Frame: 2 weeks post-treatment
Population: No data was collected/analyzed.
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: L-1 Norm Distance on Bacterial Reads (Intestinal)
Description: L-1 norm distance on bacterial reads (intestinal) from rectal swabs of 50 children. L1-norm distance on bacterial reads (intestinal) - L1 norm is equivalent to Shannon's diversity. Shannon's Alpha Diversity combines richness and diversity. Shannon's index of diversity (alpha diversity) measures both the number of species and the inequality between species abundances. A large value is given by the presence of many species with well balanced abundances.
Time Frame: 2 weeks post-treatment
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 208
Index score | 32.98 (9.37) | 43.15 (12.82)

15. Secondary Outcome: L-2 Norm Distance on Bacterial Reads (Intestinal)
Description: L-2 norm distance on bacterial reads (intestinal) from rectal swabs of 450 children. L2-norm distance on bacterial reads (intestinal) - L2 norm is equivalent to Simpson's diversity. Simpson's Alpha Diversity were obtained at Baseline and Post-treatment in this study. The minimum of Simpson's index of diversity is 0, there is no maximum. Higher Simpson's index of diversity means more diverse. There are no subscales.
Time Frame: 2 weeks post-treatment
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 208
Index score | 14.81 (5.72) | 20.46 (7.83)

16. Secondary Outcome: Changes in Normalized Reads for Campylobacter Species
Description: Reduce in normalized reads for Campylobacter species using DNA-seq from rectal swabs of 450 children.
  We compare the read numbers of Campylobacter species in each treatment group. Campylobacter is associated with disease. Reduction in Campylobacter species burden may reduce diarrhea-related mortality.
Time Frame: 2 weeks post-treatment
Measure: Number; unit: number of reads
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 208
number of reads | 1886.12 | 549.48

17. Secondary Outcome: Resistome
Description: Chao1 total resistance gene determinant richness using DNA-seq from rectal swabs of 450 children.
  We calculated Chao1 total resistance gene determinant richness across arms. Species richness is the simplest measure of biodiversity and is just a count of the number of different species in a given area.
Time Frame: 2 weeks post-treatment
Measure: Mean (Standard Deviation); unit: number of species
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 208
number of species | 3.98 (3.5) | 2.23 (2.02)

ADVERSE EVENTS:
Time Frame: 14 days following azithromycin or placebo treatment. Deaths were assessed up to 180 days post-treatment. Adverse Events were assessed 14 days following azithromycin or placebo treatment
Description: We report adverse events and clinic visits during the 2-week period immediately after treatment to better understand the safety and short-term impact of azithromycin compared with placebo in young children.
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/209
Serious Adverse Events (participants affected / at risk) | 0/221 | 0/209
Other Adverse Events (participants affected / at risk) | 44/221 | 42/209
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin (N=221) | Placebo (N=209)
Fever (self-report) (General disorders) | 37 | 42 — 14 days following azithromycin or placebo treatment among children aged 0-59 months
Abdominal pain (General disorders) | 0 | 2 — 14 days following azithromycin or placebo treatment
Vomiting (Gastrointestinal disorders) | 16 | 4 — 14 days following azithromycin or placebo treatment among children
Diarrhea (Gastrointestinal disorders) | 18 | 13
Constipation (Gastrointestinal disorders) | 1 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1 — 14 days following azithromycin or placebo treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT03676751/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03676751/SAP_001.pdf